CLINICAL TRIAL: NCT02556866
Title: Multicenter Randomized Double-blind Study Comparing the Efficacy and Safety of Rituximab in Combination With Corticosteroids to Corticosteroids Plus Placebo in the Treatment of Non-infectious Active Mixed Cryoglobulinemia Vasculitis
Brief Title: Rituximab Plus Corticosteroids in Non-infectious Active Mixed Cryoglobulinemia Vasculitis
Acronym: ESBAM
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P120122; 2013-000844-24 (EudraCT Number)
Record Dates: First submitted 2015-07-20; First posted 2015-09-22 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Cryoglobulinemia; Systemic Vasculitis
MeSH Terms: conditions — Cryoglobulinemia; Systemic Vasculitis | interventions — Rituximab; Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rituximab (Experimental): Prednisone treatment plus rituximab administered by slow intravenous infusion at 375 mg/m2 at D1, D8, D15 and D22.
  Interventions: Drug: rituximab; Drug: Prednisone
- placebo (Placebo Comparator): Prednisone treatment plus placebo administered by slow intravenous infusion at day 1 (D1), D8, D15 and D22.
  Interventions: Drug: Prednisone; Drug: Placebo

INTERVENTIONS:
Drug: rituximab — Prednisone treatment plus rituximab administered by slow intravenous infusion at 375 mg/m2 at D1, D8, D15 and D22.
  Arms: rituximab
Drug: Prednisone
Drug: Placebo
  Arms: placebo

SUMMARY:
Multicenter randomized double-blind study comparing the efficacy and safety of rituximab in combination with corticosteroids to corticosteroids plus placebo in the treatment of non-infectious active mixed cryoglobulinemia vasculitis.

DETAILED DESCRIPTION:
Cryoglobulinemia are responsible for systemic vasculitis, and the most frequently targeted organs are the skin, joints, kidneys and peripheral nervous system. Cryoglobulinemia vasculitis are associated with significant morbidity and mortality, and require therapeutic intervention. Management of non-infectious mixed cryoglobulinemia vasculitis is based on corticosteroids, plasma exchange, and/or immunosuppressants. These treatments are associated with frequent side effects. To date, no study has evaluated the efficacy and safety of these different therapeutic options, explaining the lack of recommendations.

Rituximab, a monoclonal antibody directed against CD20, has emerged as a novel therapeutic option in B-cell related disorders. Data from the French AutoImmunity and Rituximab (AIR) registry recently reported the positive effect of rituximab in non-infectious mixed cryoglobulinemia vasculitis. More recently, the multidisciplinary national French CryoVas survey also suggested a significant superiority of the combination corticosteroid plus rituximab compared to the corticosteroids alone in terms of complete clinical and immunological responses and corticosteroid sparing. However, no randomized controlled data addressing this issue has been published to date.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be at least 18 years of age or older, without any upper age limit
2. Patient informed and agreed to participate, and gave informed consent,
3. Patient with active cryoglobulinemia vasculitis define by positive cryoglobulinemia and a clinically active vasculitis with skin, joint, renal, peripheral nerve, central neurological, digestive, pulmonary and/or cardiac involvement (no histological evidence needed if presence of purpura demonstrated),
4. Patient with primary Sjögren's syndrome, systemic lupus erythematosus, or another auto-immune disease, or B-cell non-Hodgkin lymphoma (with cryoglobulinemia as the only therapeutic indication), or essential mixed cryoglobulinemia,
5. Naive or relapsing patients, without modification (initiation or increase) of immunosuppressive therapy in the month prior the inclusion,
6. For women of child bearing age: negative pregnancy test during the inclusion, and effective contraception during the period of 12 months after the latest rituximab infusion or placebo,
7. Patients with severe vasculitis must be treated in the 15 days prior inclusion by 3 bolus of methylprednisolone (15 mg/kg/d) AND 3 to 7 plasma exchanges (exchange volume of 60 ml/kg/session).

Exclusion Criteria:

1. Patient with a medium and small size vessels vasculitis unrelated to cryoglobulinemia (granulomatous with polyangiitis (Wegener's disease), microscopic polyangiitis, eosinophilic granulomatous with polyangiitis (Churg-Strauss syndrome), polyarteritis nodose, IgA vasculitis, hypersensitivity vasculitis, infectious vasculitis, hypocomplementemic urticarial vasculitis),
2. Patient with a large size vessels vasculitis,
3. Patient with non active cryoglobulinemia vasculitis,
4. Patient with immunosuppressive therapy introduced or increased in the month prior to the inclusion,
5. Patients receiving corticosteroid therapy > 0.5 mg/kg/d for more than one month before the inclusion or > 1 mg/kg/d for more than two weeks before the inclusion,
6. Patient who had received rituximab therapy within the 12 months before the inclusion,
7. Pregnancy in progress or needed , breast feeding,
8. HIV-positive status,
9. Patient with active hepatitis B or C infection,
10. HBs Ag-positive and/or HBV DNA detectable in the blood*,
11. Patients with known hypersensitivity reaction to the active substance or any of the excipients, or to murine proteins,
12. Contraindication to rituximab,
13. Active infections at screening,
14. Patient in guardianship,
15. Patient already included in a biomedical research protocol,
16. No social security scheme (Beneficiaries or eligible),
17. History of cancer during the last 3 years before inclusion, including solid tumors, hematological malignancies (except lymphoproliferative disorder associated with the mixed cryoglobulinemia vasculitis), and carcinoma in situ (except basal cell and squamous cell carcinoma of the skin that have been treated or excized and cured)"

    * If the hepatitis B core antibody (anti-HBc) is positive, the benefit/risk will be evaluated by an hepatologist before inclusion, and patient, if enrolled, will be monitored until the end of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-07-17 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Complete clinical response of vasculitis symptoms (yes-no, i.e. success-failure) with corticosteroid withdrawal (prednisone at 0 mg/day) at week (W) 24, with at least one clinical response at W4 | Week 24
  The complete clinical response is defined by the remission of all affected organs involved at baseline and the absence of clinical relapse.

SECONDARY OUTCOMES:
Partial clinical response | Week 24
  Partial clinical response defined by an improvement of at least half of organ impairments present at baseline

OTHER OUTCOMES:
Evolution of cryoglobulinemia (positive or negative) | Week 24
Evolution of C4 complement fraction (mg/L) | Week 24
Rate of early failures | Week 4
Occurrence of clinical relapse | up to Week 48
  Clinical relapse is defined by de novo appearance or reappearance of a manifestation attributable to cryoglobulinemia vasculitis during 48 weeks of follow-up,
Cumulative dose of prednisone | Week 24
quality of life | Day 1
  evolution of quality of life will be assessed by the score SF36
quality of life | Week 4
  evolution of quality of life will be assessed by the score SF36
quality of life | Week 8
  evolution of quality of life will be assessed by the score SF36
quality of life | Week 16
  evolution of quality of life will be assessed by the score SF36
quality of life | Week 24
  evolution of quality of life will be assessed by the score SF36
quality of life | Week 36
  evolution of quality of life will be assessed by the score SF36
quality of life | Week 48
  evolution of quality of life will be assessed by the score SF36
quality of life at relapse | up to Week 48
  quality of life at relapse will be assessed by the score SF36
Infusion related reactions | up to Week 4
  hypersensitivity reaction rate such as fall in blood pressure, bronchospasm, … due to rituximab or placebo infusions (included also reaction occurring after the end of infusion),
Rate of infections (severe or not) and other complications related to corticosteroids | up to Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Patrice CACOUB, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Pitié Salpetriere Hospital, Paris, France